CLINICAL TRIAL: NCT06867575
Title: Effects of Progressive Relaxation Exercises on Sleep Quality, Psychological Resilience and Quality of Life in Nursing Students: A Randomized Controlled Trial
Brief Title: Effects of Progressive Relaxation Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Assistant Professor of Nursing, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0004
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Nursing Caries; Progression; Sleep
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled trial planned to examine the effects of progressive relaxation exercises on sleep quality, psychological resilience and quality of life in nursing students.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Students will be randomly assigned (using online randomization software) to experimental and control groups. Students will know that they are participating in the study and the interventions that will be applied to them, but they will be blinded by not knowing which group they are in. The study data will be collected by a second researcher who is blinded to the groups. In the statistical analysis of the data, the groups will be labeled as group 1 and group 2, and the third researcher will be blinded when evaluating the results. Thus, the third researcher will be blinded to the study groups. In order to avoid bias in the evaluation of the results, the first researcher, who is not blinded, will not participate in any stage of the evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation group (Experimental): Progressive Relaxation Exercises
  Interventions: Other: Progressive Relaxation Exercise
- Control group (No Intervention): The students who formed the control group and accepted to participate in the study will be asked to fill out the "Descriptive Characteristics Form", "Pittsburgh Sleep Quality Index (PSQI)", "Adult Resilience Scale", and "SF-36 Quality of Life Scale" in the first meeting. After filling out the data collection tools in the first meeting in the classroom, no intervention will be made. At the end of the 4th week follow-up period, separate data collection forms and post-test results will be obtained. The control group will be given a progressive relaxation exercise audio recording and booklets with written instructions stated in the audio recording.

INTERVENTIONS:
Other: Progressive Relaxation Exercise — Progressive Relaxation Exercise Steps
  Arms: Progressive relaxation group

SUMMARY:
When the literature is examined, it is observed that the effects of progressive relaxation exercises on pain, anxiety and sleep quality have been frequently investigated in different populations. Studies conducted with nursing students focus on dysmonorrhea and clinical anxiety and stress . A limited number of studies have focused on the quality of life of students . There is no study examining the effects of progressive relaxation exercises on sleep quality, psychological endurance and quality of life together. Therefore, the aim of our study is to examine the effects of progressive relaxation exercises applied to nursing students on sleep quality, psychological endurance and quality of life. It is thought that our study results will contribute to the literature in terms of their originality.

DETAILED DESCRIPTION:
This research is a randomized controlled trial planned to examine the effects of progressive relaxation exercises on sleep quality, psychological resilience and quality of life in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a student in the Department of Nursing

  * Being willing to participate in the study
  * Not having a chronic disease that may prevent exercise (COPD, heart failure, etc.)
  * Not having a hearing problem
  * Not having a psychiatric diagnosis (major depression, anxiety disorders, etc.) and not using medication for anxiety or depression
  * Having a computer and technological devices at home
  * Being able to use a mobile phone (IOS-Android)
  * Having internet access
  * Being able to speak Turkish
  * Not having used techniques such as meditation, hypnosis, yoga for the last 6 months before the study
  * Not having a neurological, systemic, or psychiatric disease.

Exclusion Criteria:

* • Nursing students who do not volunteer to participate in the study,

  * Those who have any health problems during the application process,
  * Those who cannot continue the study for any reason,
  * Those who want to withdraw from the study with their own consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Average sleep quality score | First week, 4th week
  Pittsburgh Sleep Quality Index: This scale is a 19-item self-report scale that evaluates sleep quality and disturbances in the past month. The PSQI consists of 24 questions, 19 of which are answered by the participant, while 5 questions are answered by the spouse or roommate. The scale is divided into 7 main components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Sleep Efficiency, Sleep Disturbances, Sleep Medication Use, and Daytime Dysfunction. Each component is scored between 0 and 3, and these scores give a total result between 0 and 21. A total score above 5 indicates poor sleep quality.
Average resilience scores for Adults | First week, 4th week
  The scale containing a total of 33 items is in 5-point Likert type. The scale consists of 6 sub-dimensions. Of these, 'structural style' (3, 9, 15, 21) and 'perception of future' (2, 8, 14, 20) are measured with 4 items each; 'family harmony' (5, 11, 17, 23, 26, 32), 'self-perception' (1, 7, 13, 19, 28, 31) and 'social competence' (4, 10, 16, 22, 25, 29) are measured with 6 items each and 'social resources' (6, 12, 18, 24, 27, 30, 33) are measured with 7 items. In the scale, positive and negative features are on separate sides in order not to cause biased evaluation. Five separate boxes were created for the answers. The scoring method was left free in evaluating the level of psychological resilience as low or high. The validity and reliability Cronbach alpha coefficient of the scale was determined as 0.86 (1) by Basım and Çetin (2011), and 0.89 in this study. Considering that psychological resilience increases as the scores increase, the scoring is done as 1-2-3-4-5 from left to right
Avarage Quality of Life scores | First week, 4th week
  SF-36 Quality of Life Scale: The scale consists of 36 items and these provide the assessment of different health dimensions under 8 subscales: 1) Physical function (10 items) 2) Social function (2 items) 3) Role limitations due to physical problems (4 items) 4) Role limitations due to emotional problems (3 items) 5) Mental health (5 items) 6) Energy/vitality (4 items) 7) Pain (2 items) 8) General health perception (5 items) (Ware & Sherbourne, 1992). The scale is assessed by considering the last 4 weeks. A form evaluating the last 1 week was also applied in order to create the acute form. The assessment is made in Likert type (three-point-six-point) except for items 4 and 5; items 4 and 13 and 5 are answered in a yes/no format. Instead of giving a single total score, the scale gives a total score for each subscale separately. The second question of the scale, 'Compared to last year, how do you evaluate your health now?' only includes one-year changes, but this question is not included

CONTACTS AND LOCATIONS:
Overall Officials: Necibe DAĞCAN ŞAHİN, PhD, Principal Investigator — Kütahya Health Sciences University, Faculty of Health Sciences; Burcu NAL, PhD, Study Director — Kütahya Health Sciences University, Faculty of Health Sciences; Sema ÜSTÜNDAĞ, PhD (c), Study Director — Kütahya Health Sciences University, Faculty of Health Sciences
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No